CLINICAL TRIAL: NCT01190371
Title: Confirmation of Artemisinin Tolerance in Malaria Parasites Trial in Kilifi
Brief Title: Have Malaria Infections in Kenya Become Less Responsive to Artemisinin Treatment?
Acronym: CATMAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: University of Oxford (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEMRI_CT_2010/0013; SSC 1821 (Other: KEMRI Scientific Steering Committee)
Record Dates: First submitted 2010-08-24; First posted 2010-08-27 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2017-07

CONDITIONS: Malaria
Keywords: Artemisinin tolerance
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artesunate (Other): Confirmation of artemisinin tolerance
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Oral, once daily, 7-day regimen of artesunate 2mg/kg/day

SUMMARY:
The purpose of this study is to determine whether P. falciparum infections in Kilifi District have developed tolerance to the artemisinin class of drugs.

DETAILED DESCRIPTION:
Artemisinin-based combination therapies (ACT) are the treatment of choice for episodes of uncomplicated P. falciparum malaria in all endemic countries. Rapid clearance of pathogenic blood stage malaria parasites by artemisinins is associated with swift recovery from mild malaria and reduced mortality from severe forms of the disease. In Kenya, and most malaria endemic sub-saharan Africa, artemether-lumefantrine has been introduced as first-line treatment in the public health care sector in 2006. Alarmingly, despite the short time since the introduction of ACTs artemisinin-resistant P. falciparum malaria has already emerged in South-East Asia, an area that has historically been the cradle of global spreads of drug-resistant malaria parasites.

In a previous study in Kilifi we have observed a significant drop in early response rates to treatment with two ACTs from 2005 to 2008. Conventional markers of potential changes in anti-parasitic host immunity, drug exposure, or baseline parasite biomass could not account for the observed time-dependent change in response rates.

This protocol aims to establish with reasonable confidence whether P. falciparum infections in Kilifi District have developed tolerance to the artemisinin class of drugs. We propose to study treatment response rates to an established 7-day regimen of artesunate alone in the treatment of uncomplicated P. falciparum malaria in children aged 6 months to 10 years, at the KEMRI study site in Pingilikani, Kilifi District, Kenya. The study will also assess (i) pharmacokinetic parameters of artesunate; (ii) ex vivo and in vitro chemosensitivity of parasite isolates to DHA; (iii) genetic determinants of altered in vivo and in vitro responses to DHA; and (iv) ex vivo expression profiles in normally vs. slowly responding P. falciparum infections before and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6 months to 10 years, inclusive
* mono-infection with P. falciparum detected by microscopy;
* parasitaemia of 10,000-300,000/µl asexual forms;
* presence of axillary temperature ≥ 37.5 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* informed consent from a parent or guardian.

Exclusion Criteria:

* presence of clinical danger signs: not able to drink or breast-feed, vomiting (>twice in 24 hours), recent history of convulsions (>1 in 24h), unconscious state, unable to sit or stand;
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe acute malnutrition defined as weight for height <70% of the median NCHS/WHO (Appendix 2);
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics or pharmacodynamic assessments (e.g., antibiotics with known antimalarial activity); and
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s).

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study will be the re-infection-adjusted day 28 failure rate | Day 0-28
  Cure is defined as clearance of asexual P. falciparum parasitemia until day 7 and no recrudescence of asexual P. falciparum parasitemia until day 28. Re-infections are defined by genetic fingerprinting methods as newly emerging parasite clones during follow-up.

SECONDARY OUTCOMES:
The proportion of patients with positive malaria smears | 24hr, 48hr, 72hr
  The number of patients still having parasites at these time points divided by the total treated will give an estimate of early cure rates or estimates of early treatment failure rates as a percentage.
The percentage reduction of parasitaemia from baseline | 24hr, 48hr, 72hr
  These results will be used to compute the percentage of uncleared parasites so as to evaluate cases of early treatment failure according to the WHO criteria.
The mean time to parasite clearance | Up to day 7
  Estimated by parametric survival analysis will give an estimate of how long the drug takes to clear parasites from the time of first dosing till the time of the first negative smear.
The mean time to fever clearance | Up to day 7
  Estimated by parametric survival analysis mean time to fever clearance will be estimated to reflect the time it takes the the temperature to settle down consistently for at least 24 hours.
To estimate the rates for late clinical and parasitological failure rates | Days 28 and 42
  We will estimate the cumulative incidence of success and failure rates at days 28 and 42, by both PCR-uncorrected and PCR-corrected for recrudescence

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, Principal Investigator — KEMRI Centre for Geographic Medicine Research (Coast), University of Oxford, England; Steffen Borrmann, Principal Investigator — KEMRI Centre for Geographic Medicine Research (Coast), Heidelberg University of Medicine, Germany
Locations (3):
- Kenya (3):
  - Kadzinuni Dispensary, Kadzinuni, Kilifi County
  - Junju Dispensary, Kilifi
  - Pingilikani Dispensary, Kilifi